CLINICAL TRIAL: NCT06256341
Title: HHV-6-specific T-cell Reconstitution Among Children and Adolescents After Allogeneic Stem.
Acronym: CIRAST HHV-6
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: CIRAST HHV-6
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: allogeneic stem cell transplantation; Human herpesvirus 6 (HHV-6); T-lymphocytes; CD4+ or CD8+ T-cells

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- allogeneic HSCT peripheral blood: 3, 6, 9, 12, 18 and 24 months after allogeneic HSCT peripheral blood mononuclear cells were isolated from patient blood, stimulated with HHV-6-specific antigen (U54) and cultured for 10 days.
  Interventions: Other: Cell cultivation, Antigen testing
- healthy blood: One blood sample from a age and sex matched healthy controls without any inflammatory, immunological or infectious disease was taken. mononuclear cells were isolated from patient blood, stimulated with HHV-6-specific antigen (U54) and cultured for 10 days.
  Interventions: Other: Cell cultivation, Antigen testing

INTERVENTIONS:
Other: Cell cultivation, Antigen testing — day 10, peripheral blood mononuclear cells were re-stimulated with the virus antigen U54 for 6 hours and, thereafter, stained for surface markers (CD3, CD4, CD8, CD56) and intracytoplasmatic activation markers (IL-2, IFN-γ, TNF-α) for flow cytometric detection of virus-specific T-cells. T-cells with intracytoplasmic expression of activation markers after stimulation with the virus antigen are HHV-6-specific T-cells. This indicated HHV-6 specific cellular immunity.
  No more interventions in human except blood sampling, only basic research.

SUMMARY:
Human herpesvirus 6 (HHV-6) causes only minor symptoms in healthy individuals but in immunosuppressed patients, e.g., patients after allogeneic stem cell transplantation (HSCT), HHV-6 reactivations can lead to diseases in different organ systems. HHV-6 reactivations have also been reported to be a cause for delayed engraftment, a trigger of graft-versus-host disease and a co-factor for other virus reactivations. T-lymphocytes play an important role in the control of virus reactivations. Little is known about the development of virus-specific T-cells after allogeneic HSCT.

DETAILED DESCRIPTION:
Background:

Human herpesvirus 6 (HHV-6) causes only minor symptoms in healthy individuals but in immunosuppressed patients, e.g., patients after allogeneic stem cell transplantation (HSCT), HHV-6 reactivations can lead to diseases in different organ systems. HHV-6 reactivations have also been reported to be a cause for delayed engraftment, a trigger of graft-versus-host disease and a co-factor for other virus reactivations. T-lymphocytes play an important role in the control of virus reactivations. Little is known about the development of virus-specific T-cells after allogeneic HSCT.

Objective:

The aim of this study was the description of the HHV-6 specific cellular immunity in children and adolescents after allogeneic HSCT in the context of the clinical course.

Study design and participants:

For this prospective, cross-sectional study, 28 children and adolescents after allogeneic HSCT who received follow-up support at the respective centers were included. Patients were enrolled up to 24 months after allogeneic HSCT.. Peripheral venous blood was drawn 3, 6, 9, 12, 18, and 24 months after allogeneic HSCT. Furthermore, a blood sample was taken from 25 age- and sex-matched healthy controls without any inflammatory, immunological, or infectious diseases. This study was approved by the Institutional Review Board of the Medical University Graz and patients, parents or legal guardians of patients gave written informed consent in accordance with the Declaration of Helsinki.

Methods:

3, 6, 9, 12, 18 and 24 months after allogeneic HSCT peripheral blood mononuclear cells were isolated from patient blood, stimulated with HHV-6-specific antigen (U54) and cultured for 10 days. Furthermore, a blood sample was taken from 25 age- and sex-matched healthy controls without any inflammatory, immunological, or infectious diseases.

On day 10, peripheral blood mononuclear cells were re-stimulated with the virus antigen U54 for 6 hours and, thereafter, stained for surface markers (CD3, CD4, CD8, CD56) and intracytoplasmatic activation markers IL-2 (Interleukin-2), IFN-γ (Interferon-γ), TNF-α (tumor necrosis factor-α) for flow cytometric detection of virus-specific T-cells. T-cells with intracytoplasmic expression of activation markers after stimulation with the virus antigen are HHV-6-specific T-cells. This indicated HHV-6 specific cellular immunity.

The virus-specific immunity of patients to HHV-6 was compared to the virus-specific immunity of children and adolescents of a control group.

ELIGIBILITY:
Inclusion Criteria:

Patients who have undergone allogeneic SCT (stem cell transplantation) at one of the participating centers in the last 24 months or who will undergo allogeneic SCT during the study period (up to 3 months before the end of the study) and complete follow-up care at the respective centers

* Age> 1 year
* Written consent by participant or legal guardian

Exclusion Criteria:

* severe SCT-associated complications during the study period: Rejection of the transplant ("graft failure") severe graft-versus-host disease (GVHD grade 3 or 4)
* Relapse of the (malignant) underlying disease or occurrence of another complication (e.g. secondary malignancy), which represents an indication for cytotoxic chemotherapy (or re-transplantation) during the examination period.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 28 children with adolescent after allogeneic HSCT 25 healthy cildren as control (age and sex mached)
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2014-03-14 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
CD4+ controls | 1 day
  secretion of IL-2, IFN-γ as well as TNF-α (single cytokines and in combination) i T-cells after stimulation with the HHV-6 specific antigen U54
CD8+ patients after allogeneic HSCT | 24 month
  secretion of IL-2, IFN-γ as well as TNF-α (single cytokines and in combination) i T-cells after stimulation with the HHV-6 specific antigen U54
CD8+ controls | 1 day
  secretion of IL-2, IFN-γ as well as TNF-α (single cytokines and in combination) i T-cells after stimulation with the HHV-6 specific antigen U54
CD4+ patients after allogeneic HSCT | 24 month
  secretion of IL-2, IFN-γ as well as TNF-α (single cytokines and in combination) i T-cells after stimulation with the HHV-6 specific antigen U54 of IL-2, IFN-γ as well as TNF-α (single cytokines and in combination) in both

IPD SHARING:
Plan to Share IPD: Undecided